CLINICAL TRIAL: NCT03232112
Title: Does Glucagon-like Peptide (GLP-1) Receptor Agonist Stimulation Reduce Alcohol Intake in Patients With Alcohol Dependence?
Brief Title: Does Treatment With GLP-1 Reduce Alcohol Intake in Patients With Alcohol Dependence?
Acronym: EXALT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anders Fink-Jensen, MD, DMSci (Other)
Collaborators: The Novavì outpatient clinics, Copenhagen (Unknown); Rigshospitalet, Denmark (Other); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Anders Fink-Jensen, MD, DMSci, Professor, MD, DMSci, Psychiatric Centre Rigshospitalet
Organization: Psychiatric Centre Rigshospitalet (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EXALT study
Record Dates: First submitted 2017-07-20; First posted 2017-07-27 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Alcohol Dependence, in Remission; Addiction, Alcohol
Keywords: Alcohol; Addiction; Glucagon Like Peptide-1; GLP-1
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — Exenatide; Injections; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, placebo-controlled.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: An un-blinded nurse will be responsible for carrying out the randomization of the patients in REDCap. When randomization is carried out, the nurse will ensure that the patient gets the treatment that he/she is allocated to. Patients, investigators, other care givers performing assessments and persons performing data analysis will remain blinded from the time of randomization until time of database unlock. In order to maintain the blinding of the patients, the nurse will prepare the injection in a separate room and the patients will be blindfolded as the injection is given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exenatide 2 MG Injection (Active Comparator): Bydureon® (exenatide) is supplied as powder and solvent for prolonged release injection (once-weekly). Bydureon® is delivered in a carton containing four pens. Each single-dose, dual-chamber pen contains 0.65 ml of diluent and 2 mg of exenatide, which are isolated until mixed by the person administering the drug. Needles are supplied with the pen.
  Interventions: Drug: Exenatide 2 MG Injection
- BD PosiFlush (saline) (Placebo Comparator): The placebo will be supplied for as pre-filled saline syringes (BD PosiFlush™, BD Worldwide) containing 3 ml each. Needles are bought separately.
  Interventions: Drug: BD PosiFlush (saline)

INTERVENTIONS:
Drug: Exenatide 2 MG Injection — Subcutaneous injection once-weekly
  Other Names: Bydureon Pen, 2 Mg, Extended Release
  Arms: Exenatide 2 MG Injection
Drug: BD PosiFlush (saline) — Subcutaneous injection once-weekly
  Other Names: Saline
  Arms: BD PosiFlush (saline)

SUMMARY:
The study is a double-blinded, randomized, placebo-controlled, 26-weeks clinical trial. The objective of the trial is to investigate the effects of the GLP-1 receptor agonist Bydureon® (exenatide) vs. placebo on alcohol intake in patients with a diagnosis of alcohol dependence.

DETAILED DESCRIPTION:
Number of patients and target population:

144 patients with a diagnosis of alcohol dependence and 25 healthy participants (described later).

The patients included in the trial will be treated for 26 weeks with once-weekly subcutaneous injection of Bydureon® (exenatide) 2 mg or placebo. The medication will be provided as a supplement to a standard, psychosocial alcohol treatment program. There will be a long-term follow up 26 weeks after end of participation in the trial

Recruitment of the patients:

The patients will be recruited from the out-patient treatment clinics "Novavì ambulatorierne" in suburbs of Copenhagen. All patients will receive psychosocial alcohol treatment based on psycho educative elements, motivational interviewing and cognitive behavioural treatment. Skilled staff members administer the treatment.

The recruitment procedure starts when the patients contact Novavì ambulatorierne. The first contact is often without any appointment - i.e. as "drop-in". At this point the patients will be met by a healthcare provider at his/her local Novavì ambulatorie. The healthcare provider will be a nurse or a doctor. The patient will be treated in accordance to the Novavì guidelines, i.e. start of abstinence treatment and a plan will be agreed on. At this point, the health personal will also ask if the patient could be interested in our project. Information regarding the project will also be available on the web page of Novavì. If he/she is interested and the patient fits the inclusion criteria the patient will be handed written information about the trial, and an information meeting will be set up a few days later. The patient will be informed about his/her right to bring a friend or adviser.

Pre-treatment evaluation/screening:

Before screening, all patients will be provided with oral and written information about the trial, including the most common adverse events, and the procedures involved in the study. All patients will be fully in-formed, verbally and in writing, of their rights and responsibilities while participating in the trial. Screening examinations will only be performed after the patient has agreed to participate and has signed and dated the informed consent form.

Screening:

At screening examinations, the patient will be asked about his/her alcohol intake the previous 30 days. The information will be recorded via TLFB (Time Line Follow Back) method. The patient will be asked questions about his/her lifetime alcohol consumption, previous treatment and general information about psychosocial factors, i.e. education level, employment and marital status.

In addition, Alcohol Users Identification Test (AUDIT) score, the Clinical Institute Withdrawal Assessment of Alcohol Scale Revised (CIWA-Ar), The Drug User Identification Test (DUDIT) score, Major Depression Inventory (MDI) score (related to the SPECT results), Penn alcohol craving scale (PACS), smoking status (Fagerströms test), height, weight, waist circumference, blood pressure and pulse will be registered. In order to evaluate psychosocial status a general assessment including questionnaires regarding health (SF-36), Symptom checklist (SCL-92) and Screen for Cognitive Impairment in Psychiatry (SCIP) - test will be performed.The patients will also be asked questions regarding somatic symptoms, i.e. GI-symptoms, in order to obtain baseline information. In addition, other medications than Bydureon® will be registered.

Different safety blood samples and a urine test will be collected. A blood sample and a urine sample will be saved for an investigational biobank and a biobank for future research.

Weekly visits:

The patient will meet every week to get his/her weekly injection by the un-blinded nurse. The nurse will collect a weekly alcohol diary and hand them a new one, for the following week.

Examinations during and in the end of the trial:

At week 4, 12 and 20, parts of the baseline examinations - including blood samples - will be conducted. The alcohol diaries collected in relation to the weekly injection-visits will be used as template for the 30 day TLFB at the examinations, i.e. the examiner will fill out the TLFB based on the diaries and in close collaboration with the patient. At week 26, the final examination will take place repeating all the baseline examinations.

Long-term follow up 26 weeks after end of participation in the trial:

All participants completing the final week 26 examination, will be contacted after six months, and invited to a follow up meeting . TLFB, PACS, AUDIT and Fagerstrøms questionnaire will be repeated. A new questionnaire, which gives us a better characteristic of the patient's alcohol history, "Alco-life" will be registered. A single blood test, (PEth) will be collected.

Study of the possible neuro molecular and -anatomical underpinnings:

In addition to the clinical outcome parameters, the investigators will explore the neuro molecular and -anatomical underpinnings of potential therapeutic effects of Bydureon® in two subgroups of patients who are treated with either Bydureon® or placebo. In order to study this,two different brain scans will be performed: Single-photon emission computed tomography (SPECT)-scan (sixty) and functional Magnetic Resonance Imaging (fMRI)-scan (seventy-five patients) at baseline and after 26 weeks of treatment. The patients will be included continuously until the aimed number (i.e. sixty and seventy-five patients for each scan type, respectively) have completed base line scan. The patients will be asked to undergo both scan types (except from the last fifteen patients out of the seventy-five patients included for scans, who will only undergo fMRI scan) as the information from both scans will be paired during evaluation. When baseline scans are performed, the patients start the treatment they were randomized for at inclusion.

The SPECT-scan:

Studies have lately reported on a GLP-1-induced upregulation of the rat dopamine transporter activity in vitro. In the present study, the investigators want to investigate whereas GLP-1 receptor stimulation induces changes in the striatal dopamine transporter availability in humans. The investigators will conduct the SPECT brain scan with the dopamine transporter ligand 123I-2-b-carbomethoxy-3b-(4-iodophenyl)-N-(3-fluoropropyl) nortropane ([123I]-FP-CIT) (DaTSCAN, Amersham Health). The SPECT scans will be conducted at the Neurobiology Research Unit, Rigshospitalet.

The fMRI-scan:

The fMRI-scan measures brain blood flow, which reflects activity in different areas of the brain. We will test two different paradigms: 1) Alcohol cue sensitivity. Sixty alcohol-related and 45 neutral stimuli are presented using a block design. Following each block, the patients rate the intensity of their alcohol craving on a visual analogue scale ranging from 0 (no craving) to 100 (extremely extensive craving). 2) Spatial working memory. Spatial working memory is assessed using 2-back and 0-back variants of the N-back task for the active working memory and control conditions.

Study-schedule for the 25 healthy fMRI-participants:

To have comparable standard data in the fMRI alcohol related paradigm, 25 healthy participants with no record of alcohol dependence will be recruited. The participants will be matched with gender and age of the patients and have to fulfil the exclusion-criteria.

Day 1: The participants will have an interview about physical symptoms, diagnosis and current medication. They will be asked to fill out the Alcohol Users Identification Test (AUDIT), the Drug Users Identification Test (DUDIT), have a basic physical examination and a blood and a urine test done.

Day 2: They will start with the Screen for Cognitive Impairment in Psychiatry (SCIP) test, and afterwards have the fMRI scan done.

ELIGIBILITY:
Inclusion Criteria:

* Informed oral and written consent
* Diagnosed with alcohol dependence according to the criteria of International Classification of Diseases (ICD) 10, World Health Organization and DSM-5
* Alcohol use disorder identification test (AUDIT) score >15
* Age 18 - 70 years
* Heavy alcohol drinking defined as having alcohol consumption over 60 g of alcohol per day (men) or 48 g of alcohol per day (women) for at least 5 days in the past 30 days prior to inclusion measured by the TLFB method.

Exclusion Criteria:

* Severe psychiatric disease, defined as a diagnosis of schizophrenia, paranoid psychosis, bipolar dis-order or mental retardation
* A history of delirium tremens or alcohol withdrawal seizures
* No serious withdrawal symptoms at inclusion (a score higher than 9 on the Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised (CIWA-Ar)) at baseline examinations
* Present or former neurological disease including traumatic brain injury
* Present or former diagnosis of type 1 or type 2 diabetes or plasma Haemoglobin A1c (HbA1c ) ≥48 moll/L at inclusion
* Females of child bearing potential who are pregnant, breast-feeding or have intention of becoming pregnant within the next 9 months (26 weeks plus three months after discontinuation of Bydureon®) , or are not using contraceptives (during the whole study period) considered as highly effective (combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable) intrauterine device - IUD, IUS, bilateral tubal occlusion, vasectomised partner, sexual abstinence) (33)
* Pregnancy (serum hCG > 3 at inclusion) Impaired hepatic function (liver transaminases >3 times up-per normal limit)
* Impaired renal function (eGFR < 50 ml/min and/or microalbuminuria) Impaired pancreatic function (any history of acute or chronic pancreatitis and/or amylase > 2 times upper limit)
* S-triglycerides > 10 mmol/l
* Former medullary thyroid carcinoma (MTC) and/or family history with MTC and/or Multiple Endo-crine Neoplasia syndrome type 2 (MEN 2)
* Cardiac problems defined as decompensated heart failure (NYHA class III or IV), unstable angina pectoris and/or myocardial infarction within the last 12 months
* Uncontrolled hypertension (systolic blood pressure >180 mmHg, diastolic blood pressure >110 mmHg)
* Concomitant pharmacotherapy against alcohol dependence including disulfiram, naltrexone, acamprosate and nalmefene or treatment with any of these compounds within 1 month prior to inclusion
* Concomitant pharmacotherapy with dopamine active drugs, such as some types of Attention Deficit Hyperactivity Disorder (ADHD) medication (methylphenidate)
* Receiving any investigational drug within the last 3 months
* Use of weight-lowering pharmacotherapy within the preceding 3 month
* Any other active substance use defined as a DUDIT-score > 6 (for men) >2 (for women) and fulfilling the criteria's for dependence of the substance according to the criteria of International Classification of Diseases (ICD) 10 (except nicotine)
* BMI <18.5 kg/m2
* Hypersensitivity to the active substance or to any of the excipients
* Only for patients undergoing brain scans: Contraindications for undergoing an fMRI scan (magnetic implants, pacemaker, claustrophobia etc.). Contraindications for undergoing a SPECT-scan (allergy towards iodine, radiation exposure, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 10 mSv in the last 12 months)
* Unable to speak and/or understand Danish
* Any condition that the investigator feels would interfere with trial participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Heavy drinking days | 30 days prior to baseline and 30 days prior to final follow up at 26 weeks
  Percent reduction in alcohol consumption, defined as total number of heavy drinking days (as days with an excess intake of 60/48 grams of alcohol per day (men and women, respectively)) for the past 30 days. This will be registered via the Timeline-Follow-Back (TLFB) method.

SECONDARY OUTCOMES:
Total alcohol consumption | 30 days prior to baseline and 30 days prior to final follow up at 26 weeks
  Percent reduction in alcohol consumption, defined as "x" grams of alcohol for the past 30 days. This will be registered via the Timeline-Follow-Back (TLFB) method.
Penn Alcohol Craving Scale (PACS) score | Baseline and 26 weeks
  Score for measuring alcohol craving
Alcohol Use Disorders Identification Test (AUDIT) score | Baseline and 26 weeks
  Screening for excessive drinking
Drug Use Disorders Identification Test (DUDIT) score | Baseline and 26 weeks
  A parallel instrument to the AUDIT for identification of individuals with drug-related problems
Screen For Cognitive Impairment in Psychiatry (SCIP) test | Baseline, 4 weeks and 26 weeks
  The 20 minute test is a simple scale developed for screening cognitive deficits
Plasma-gamma-glutamyltransferase (GGT) | Baseline and 26 weeks
  Liver parameter
Plasma-alanine aminotransferase (ALAT) | Baseline and 26 weeks
  Liver parameter
Plasma-phosphatidylethanol (PEth) | Baseline, 4, 12, 20 and 26 weeks
  Biomarker for alcohol consumption
Blood-mean cell volume | Baseline and 26 weeks
  Measure of the average volume of a red blood cell
Body weight | Baseline, 4, 12, 20 and 26 weeks
  Body weight in kilograms
Blood pressure | Baseline, 4, 12, 20 and 26 weeks
  Systolic and diastolic blood pressure
Pulse | Baseline, 4, 12, 20 and 26 weeks
  Number of heartbeats pr. minute
Waist circumference | Baseline, 4, 12, 20 and 26 weeks
  Widest abdominal circumference in centimeters
Plasma-glycemic control parameters | Baseline and 26 weeks
  HbA1c, cholesterol, triglycerides, high-density lipoprotein (HDL), low-density lipoprotein (LDL).
Kidney function | Baseline and 26 weeks (eGFR also at week 12)
  e-GFR, urine albumine/creatinine-ratio.
Short Form Health Survey (SF-36) | Baseline and 26 weeks
  36-item, patient-reported survey of patient health
Plasma amylase | Baseline and 26 weeks
  Safety (i.e. pancreatic function)
Symptom Checklist (SCL-92) | Baseline and 26 weeks
  92-item, patient-reported survey of a broad range of psychological problems and symptoms of psychopathology.
Single-photon emission computed tomography (SPECT) | Baseline and 26 weeks
  In this study we want to investigate whereas GLP-1 receptor stimulation induces changes in the striatal dopamine transporter availability in humans.
fMRI (functional magnetic resonance imaging) | Baseline and 26 weeks
  In this study we want to investigate whereas GLP-1 treatment modulate neural responses in reward processing regions including nucleus accumbens. Data from the 25 healthy participants will be used as comparable standard when analyzing the data.

CONTACTS AND LOCATIONS:
Overall Officials: Signe W. Düring, MD, Principal Investigator — The Novavi outpatient clinics, Copenhagen
Locations (1):
- Novavì ambulatorierne, Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
At the start and at the end of the study a blood sample (9ml) and a urine sample (7.2ml) will be stored in a biobank for future research. The patients will be asked to give a separate written consent. Using this biobank in the future will require a new approval from the Danish Data Protection Agency.

REFERENCES:
- [Derived] Klausen MK, Jensen ME, Moller M, Le Dous N, Jensen AO, Zeeman VA, Johannsen CF, Lee A, Thomsen GK, Macoveanu J, Fisher PM, Gillum MP, Jorgensen NR, Bergmann ML, Enghusen Poulsen H, Becker U, Holst JJ, Benveniste H, Volkow ND, Vollstadt-Klein S, Miskowiak KW, Ekstrom CT, Knudsen GM, Vilsboll T, Fink-Jensen A. Exenatide once weekly for alcohol use disorder investigated in a randomized, placebo-controlled clinical trial. JCI Insight. 2022 Oct 10;7(19):e159863. doi: 10.1172/jci.insight.159863. PMID 36066977

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT03232112/SAP_000.pdf